CLINICAL TRIAL: NCT04233034
Title: Hybrid Closed Loop Therapy and Verapamil for Beta Cell Preservation in New Onset Type 1 Diabetes (CLVer)
Brief Title: Hybrid Closed Loop Therapy and Verapamil for Beta Cell Preservation in New Onset Type 1 Diabetes
Acronym: CLVer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); University of Minnesota (Other); DexCom, Inc. (Industry); Medtronic (Industry); Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: CLVer
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Type1 Diabetes
Keywords: new onset; verapamil; hybrid closed loop; hcl; beta cell; diabetes; children; T1D; c-peptide; pediatric
MeSH Terms: conditions — Leukemia, Hairy Cell; Diabetes Mellitus | interventions — Verapamil; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- HCL and placebo (Active Comparator): Participants assigned to HCL group will initially be randomly assigned 1:1 to use either the Tandem t:slim X2 with Control-IQ technology or a Medtronic HCL system (Medtronic 670G 4.0 AHCL (prior to protocol version 5.0) or Medtronic 780G (starting with protocol version 5.0)). This group will receive intensive diabetes management with frequent contacts by study staff with the goal of near-normalization of glucose concentrations.
  Placebo will be taken orally once per day by participants in Cohort A. A dosing scheme will be followed, using 120mg tablets or 60mg half tablets.
  Whether drug is active or placebo is blinded to both participant and site.
  [Cohort B participants will not receive study drug. Instead, they will be randomized 2:1 to HCL or non-HCL.]
  Interventions: Device: HCL; Drug: placebo
- HCL and verapamil (Active Comparator): Participants assigned to HCL group will initially be randomly assigned 1:1 to use either the Tandem t:slim X2 with Control-IQ technology or a Medtronic HCL system (Medtronic 670G 4.0 AHCL (prior to protocol version 5.0) or Medtronic 780G (starting with protocol version 5.0)). This group will receive intensive diabetes management with frequent contacts by study staff with the goal of near-normalization of glucose concentrations.
  Verapamil will be taken orally once per day by participants in Cohort A. A dosing scheme will be followed, using 120mg tablets or 60mg half tablets.
  Whether drug is active or placebo is blinded to both participant and site.
  [Cohort B participants will not receive study drug. Instead, they will be randomized 2:1 to HCL or non-HCL.]
  Interventions: Device: HCL; Drug: verapamil 120mg tablet
- non-HCL and verapamil (Active Comparator): Participants assigned to non-HCL will receive a Dexcom G6 CGM and diabetes management will follow usual care by their personal diabetes health care provider.
  Verapamil will be taken orally once per day by participants in Cohort A. A dosing scheme will be followed, using 120mg tablets or 60mg half tablets.
  Whether drug is active or placebo is blinded to both participant and site.
  [Cohort B participants will not receive study drug. Instead, they will be randomized 2:1 to HCL or non-HCL.]
  Interventions: Drug: verapamil 120mg tablet; Device: non-HCL
- non-HCL and placebo (Placebo Comparator): Participants assigned to non-HCL will receive a Dexcom G6 CGM and diabetes management will follow usual care by their personal diabetes health care provider.
  Placebo will be taken orally once per day by participants in Cohort A. A dosing scheme will be followed, using 120mg tablets or 60mg half tablets.
  Whether drug is active or placebo is blinded to both participant and site.
  [Cohort B participants will not receive study drug. Instead, they will be randomized 2:1 to HCL or non-HCL.]
  Interventions: Device: non-HCL; Drug: placebo

INTERVENTIONS:
Device: HCL — Hybrid Closed Loop therapy
  Arms: HCL and placebo; HCL and verapamil
Drug: verapamil 120mg tablet — verapamil tablet
  Arms: HCL and verapamil; non-HCL and verapamil
Device: non-HCL — Usual diabetes care
  Arms: non-HCL and placebo; non-HCL and verapamil
Drug: placebo — placebo pill manufactured to mimic verapamil 120mg tablet
  Arms: HCL and placebo; non-HCL and placebo

SUMMARY:
Randomized trial of youth aged 7-<18 years with newly diagnosed stage 3 type 1 diabetes (T1D) to assess the effect of both (1) near-normalization of glucose concentrations achieved through use of a hybrid closed loop (HCL) system and (2) verapamil on preservation of β-cell function 12 months after diagnosis. Participants with body weight ≥30 kg (Cohort A) will be randomly assigned in a factorial design to (1) HCL plus intensive diabetes management or usual care with no HCL and (2) verapamil or placebo. Participants with body weight <30 kg (Cohort B) will be randomly assigned 2:1 in a parallel group design to HCL plus intensive diabetes management or to usual care with no HCL.

DETAILED DESCRIPTION:
After informed consent is obtained, potential participants will be assessed for eligibility, including eliciting medical history, physical examination, and laboratory testing (including HbA1c, auto-antibody measurement [unless positive auto-antibody results already available], and pregnancy test for females with childbearing potential).

Participants who already have positive auto-antibodies can be randomized immediately. All other participants will be scheduled for a randomization visit after the auto-antibody results are available; positive auto-antibodies are required for randomization.

Eligible participants with body weight ≥30 kg (Cohort A) will be randomly assigned to one of 4 groups: HCL and placebo, HCL and verapamil, non-HCL and placebo or non-HCL and verapamil. Eligible individuals with body weight <30 kg (Cohort B) will be randomly assigned 2:1 to either HCL or non-HCL. Randomization schedules will be separate for Cohort A and Cohort B and will be stratified by site.

Participants assigned to HCL will receive intensive diabetes management with frequent contacts by study staff with the goal of near-normalization of glucose concentrations.

Participants assigned to non-HCL will receive a Dexcom G6 continuous glucose monitor (CGM) and diabetes management will follow usual care by their personal diabetes health care provider.

Participants will be followed for 12 months from diagnosis, completing a 6 week visit timed from randomization and 13, 26, 39, and 52 week visits timed from diagnosis. Participants will have a MMTT performed, HbA1c measured, and blood drawn for mechanistic studies at Randomization, 13, 26, 39 and 52 weeks. At all follow-up visits, a physical exam will be performed, pregnancy testing performed (if indicated), insulin dose (units/kg/day) recorded, and device data downloaded.

Safety assessments will be made throughout the study by querying about episodes of severe hypoglycemia and DKA, and overall health.

Participants already enrolled in the study and using the Medtronic 670G 4.0 AHCL may transition to the Medtronic 780G if desired. Contacts will be performed to review CareLink data and check for adverse events and device deficiencies on days 1, 3 and 5 after transition from 670G 4.0 AHCL to 780G.

Prior to the 780G system becoming commercially available, study participants using the Medtronic system at 52 weeks will have the opportunity to continue using the 780G system at home until the system is commercially available OR until the CLVer trial is complete (last participant's 52-week visit), whichever comes first.

Additional Procedures for Cohort A:

Drug will be double blinded. Drug dose will be weight-dependent and will be escalated at 2-4 week intervals, up to a weight-dependent maximum if tolerated. Cohort A will have additional safety visits 1 week after initiation of study drug and after each study drug dose increase, to test blood pressure and pulse.

Local lab measurement of aspartate aminotransferase/alanine aminotransferase (AST/ALT) and creatinine will occur, and an EKG will be performed at Screening, 6, 26, and 52 weeks. Over the course of the trial, study drug dose may be decreased or discontinued if side effects occur.

ELIGIBILITY:
* Participant Inclusion Criteria:

  1. New-onset stage 3 T1D within 21 days of diagnosis (timed from start of insulin therapy), with ability to be randomized within 31 days of diagnosis (time from diagnosis to screening can be longer provided all screening testing can be completed within 31 days of diagnosis)
  2. At least one positive type 1 diabetes auto-antibody
  3. Age 7 - <18 years at the time of enrollment
  4. Willing to have a parent or legal guardian provide informed consent and child assent
  5. In a female participant with childbearing potential, not currently pregnant and willing to avoid pregnancy and breastfeeding and undergo pregnancy testing throughout the study
  6. English speaking/reading
  7. Able to swallow pills (tested with an inert imitation tablet in clinic prior to randomization)
  8. Willing to not use any non-insulin glucose-lowering agents
  9. Willing to use an insulin approved for the pump (if assigned to HCL)
  10. Willing to avoid medications containing acetaminophen, and no contraindications for ibuprofen use (in case assigned to Medtronic HCL system)
* Participant Exclusion Criteria:

  1. Ongoing use of medications known to influence glucose tolerance such as systemic steroids
  2. Other systemic disease which in the opinion of the investigator precludes participation (including psychiatric illness)
  3. Unwilling to abstain from use of HCL therapy for 12 months

     a. Personal pump and CGM use, including systems with a "suspend-before-low" function, will be allowed for participants randomized to non-HCL groups
  4. "Silent" diabetes-i.e., Stage 3 diabetes that is identified by routine oral glucose tolerance testing (OGTT) or in the course of surveillance studies but is not accompanied by fasting hyperglycemia or classic symptoms of diabetes
  5. Participation in another research study that involves diabetes care
* Additional exclusion criteria for Cohort A:

  1. Blood pressure (either systolic or diastolic) <5th percentile for age, gender, and height on two out of three measurements
  2. Pulse <2nd percentile for age and gender on two out of three measurements
  3. History of vasovagal syncopal episodes related to hypotension
  4. Abnormal EKG rhythm unless cleared for study participation by a cardiologist
  5. Underlying cardiac disease (ex. left ventricular dysfunction, hypertrophic cardiomyopathy), certain arrhythmias (ex. Atrioventricular block (AV) block, accessory pathway such as Wolff-Parkinson-White or Lown-Ganong-Levine syndromes), known liver dysfunction, known renal impairment, Duchenne's muscular dystrophy, active Graves disease or hyperthyroidism, and untreated hypothyroidism
  6. Estimated glomerular filtration rate (eGFR) < 90
  7. AST and/or ALT greater than 1.5 times the upper limit of normal
  8. Need to use of any of the following medications during the study: beta blocker, seizure medication (carbamazepine, phenobarbital, phenytoin), other antihypertensive medications, HMG-CoA reductase inhibitors, lithium, theophylline, clonidine, or aspirin
  9. Any known hypersensitivity reaction to Verapamil

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Moran, MD, Study Chair — University of Minnesota; Gregory Forlenza, MD, Study Chair — Barbara Davis Center
Locations (6):
- United States (6):
  - Stanford University, Palo Alto, California
  - Barbara Davis Center, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Indiana University, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri

REFERENCES:
- [Derived] Ekhlaspour L, Buckingham B, Bauza C, Clements M, Forlenza GP, Neyman A, Norlander L, Schamberger M, Sherr JL, Bailey R, Beck RW, Kollman C, Beasley S, Cobry E, DiMeglio LA, Paprocki E, Van Name M, Moran A; CLVer Study Group. Safety and prescribing recommendations for verapamil in newly diagnosed pediatric type 1 diabetes (T1D): The CLVer experience. J Clin Transl Endocrinol. 2024 May 18;36:100352. doi: 10.1016/j.jcte.2024.100352. eCollection 2024 Jun. PMID 38860154
- [Derived] Forlenza GP, McVean J, Beck RW, Bauza C, Bailey R, Buckingham B, DiMeglio LA, Sherr JL, Clements M, Neyman A, Evans-Molina C, Sims EK, Messer LH, Ekhlaspour L, McDonough R, Van Name M, Rojas D, Beasley S, DuBose S, Kollman C, Moran A; CLVer Study Group. Effect of Verapamil on Pancreatic Beta Cell Function in Newly Diagnosed Pediatric Type 1 Diabetes: A Randomized Clinical Trial. JAMA. 2023 Mar 28;329(12):990-999. doi: 10.1001/jama.2023.2064. PMID 36826844
- [Derived] McVean J, Forlenza GP, Beck RW, Bauza C, Bailey R, Buckingham B, DiMeglio LA, Sherr JL, Clements M, Neyman A, Evans-Molina C, Sims EK, Messer LH, Ekhlaspour L, McDonough R, Van Name M, Rojas D, Beasley S, DuBose S, Kollman C, Moran A; CLVer Study Group. Effect of Tight Glycemic Control on Pancreatic Beta Cell Function in Newly Diagnosed Pediatric Type 1 Diabetes: A Randomized Clinical Trial. JAMA. 2023 Mar 28;329(12):980-989. doi: 10.1001/jama.2023.2063. PMID 36826834

RESULTS

PARTICIPANT FLOW:
Groups:
- HCL and Placebo: Participants assigned to HCL group will initially be randomly assigned 1:1 to use either the Tandem t:slim X2 with Control-IQ technology or a Medtronic HCL system (Medtronic 670G 4.0 AHCL (prior to protocol version 5.0) or Medtronic 780G (starting with protocol version 5.0)). This group will receive intensive diabetes management with frequent contacts by study staff with the goal of near-normalization of glucose concentrations.
  Placebo will be taken orally once per day by participants in Cohort A. A dosing scheme will be followed, using 120mg tablets or 60mg half tablets.
  Whether drug is active or placebo is blinded to both participant and site.
  [Cohort B participants will not receive study drug. Instead, they will be randomized 2:1 to HCL or non-HCL.]
  HCL: Hybrid Closed Loop therapy
  placebo: placebo pill manufactured to mimic verapamil 120mg tablet
- HCL and Verapamil: Participants assigned to HCL group will initially be randomly assigned 1:1 to use either the Tandem t:slim X2 with Control-IQ technology or a Medtronic HCL system (Medtronic 670G 4.0 AHCL (prior to protocol version 5.0) or Medtronic 780G (starting with protocol version 5.0)). This group will receive intensive diabetes management with frequent contacts by study staff with the goal of near-normalization of glucose concentrations.
  Verapamil will be taken orally once per day by participants in Cohort A. A dosing scheme will be followed, using 120mg tablets or 60mg half tablets.
  Whether drug is active or placebo is blinded to both participant and site.
  [Cohort B participants will not receive study drug. Instead, they will be randomized 2:1 to HCL or non-HCL.]
  HCL: Hybrid Closed Loop therapy
  verapamil 120mg tablet: verapamil tablet
- Non-HCL and Verapamil: Participants assigned to non-HCL will receive a Dexcom G6 CGM and diabetes management will follow usual care by their personal diabetes health care provider.
  Verapamil will be taken orally once per day by participants in Cohort A. A dosing scheme will be followed, using 120mg tablets or 60mg half tablets.
  Whether drug is active or placebo is blinded to both participant and site.
  [Cohort B participants will not receive study drug. Instead, they will be randomized 2:1 to HCL or non-HCL.]
  verapamil 120mg tablet: verapamil tablet
  non-HCL: Usual diabetes care
- Non-HCL and Placebo: Participants assigned to non-HCL will receive a Dexcom G6 CGM and diabetes management will follow usual care by their personal diabetes health care provider.
  Placebo will be taken orally once per day by participants in Cohort A. A dosing scheme will be followed, using 120mg tablets or 60mg half tablets.
  Whether drug is active or placebo is blinded to both participant and site.
  [Cohort B participants will not receive study drug. Instead, they will be randomized 2:1 to HCL or non-HCL.]
  non-HCL: Usual diabetes care
  placebo: placebo pill manufactured to mimic verapamil 120mg tablet
- HCL Only: Participants weighing <30 kg at study enrollment were randomly assigned 2:1 in a parallel group design to HCL plus intensive diabetes care or usual care with no HCL.
  Participants assigned to HCL group will initially be randomly assigned 1:1 to use either the Tandem t:slim X2 with Control-IQ technology or a Medtronic HCL system (Medtronic 670G 4.0 AHCL (prior to protocol version 5.0) or Medtronic 780G (starting with protocol version 5.0)). This group will receive intensive diabetes management with frequent contacts by study staff with the goal of near-normalization of glucose concentrations.
  HCL: Hybrid Closed Loop Therapy
- Non-HCL Only: Participants weighing <30 kg at study enrollment were randomly assigned 2:1 in a parallel group design to HCL plus intensive diabetes care or usual care with no HCL.
  Participants assigned to non-HCL will receive a Dexcom G6 CGM and diabetes management will follow usual care by their personal diabetes health care provider.
  non-HCL: Usual diabetes care
Period: Overall Study
Arm/Group | HCL and Placebo | HCL and Verapamil | Non-HCL and Verapamil | Non-HCL and Placebo | HCL Only | Non-HCL Only
Started | 20 | 22 | 25 | 21 | 19 | 6
Completed | 20 | 21 | 23 | 19 | 19 | 6
Not Completed | 0 | 1 | 2 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HCL and Verapamil | HCL and Placebo | Non-HCL and Verapamil | Non-HCL and Placebo | HCL Only | Non-HCL Only | Total
Number analyzed (Participants) | 22 | 20 | 25 | 21 | 19 | 6 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 13 (3) | 12 (2) | 13 (3) | 13 (2) | 8 (1) | 9 (1) | 12 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 12 | 7 | 10 | 3 | 49
  Male | 14 | 11 | 13 | 14 | 9 | 3 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 16 | 14 | 20 | 15 | 15 | 6 | 86
  Race/Ethnicity: Black/African American | 1 | 1 | 1 | 0 | 1 | 0 | 4
  Race/Ethnicity: Hispanic | 4 | 2 | 4 | 4 | 1 | 0 | 15
  Race/Ethnicity: Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Race/Ethnicity: American Indian/Alaskan Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Race/Ethnicity: More than One | 0 | 2 | 0 | 2 | 2 | 0 | 6
Annual Household Income [Count of Participants; unit: Participants]
  <$50,000 | 5 | 3 | 5 | 2 | 2 | 0 | 17
  $50,000-<$100,000 | 5 | 3 | 4 | 6 | 5 | 3 | 26
  >=$100,000 | 12 | 12 | 15 | 8 | 12 | 3 | 62
  Missing | 0 | 2 | 1 | 5 | 0 | 0 | 8
Highest Parental Education [Count of Participants; unit: Participants]
  Less than Bachelor's | 6 | 7 | 6 | 6 | 2 | 1 | 28
  Bachelor's | 10 | 6 | 11 | 10 | 8 | 3 | 48
  Advanced Degree | 6 | 7 | 8 | 5 | 9 | 2 | 37
Health Insurance [Count of Participants; unit: Participants]
  Private | 16 | 19 | 22 | 18 | 14 | 3 | 92
  Public | 4 | 1 | 3 | 3 | 5 | 2 | 18
  None | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Missing | 0 | 0 | 0 | 0 | 0 | 1 | 1
BMI Percentile at Randomization [Median (Inter-Quartile Range); unit: Percentile] — Population: 1 participant in the Non-HCL placebo group was missing BMI percentile at randomization.
  Percentile
    number analyzed (Participants) | 22 | 20 | 25 | 20 | 19 | 6 | 112
    (all) | 78 [34 to 90] | 53 [21 to 86] | 58 [33 to 89] | 65 [37 to 80] | 43 [22 to 47] | 32 [26 to 37] | 56 [28 to 85]
Time Since Diagnosis at Randomization (days) [Mean (Standard Deviation); unit: Days] | 24 (5) | 24 (5) | 24 (5) | 25 (4) | 23 (5) | 23 (5) | 24 (5)
Lab HbA1c at Randomization (%) [Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin] — Population: 1 participant randomized to HCL + Placebo and 1 participant randomized to Non-HCL + Placebo were missing HbA1c at randomization.
  Percentage of glycosylated hemoglobin
    number analyzed (Participants) | 22 | 19 | 25 | 20 | 19 | 6 | 111
    (all) | 10.1 (1.6) | 10.3 (1.1) | 10.6 (1.7) | 10.1 (1.4) | 10.6 (1.2) | 9.4 (1.5) | 10.6 (1.7)
Systolic Blood Pressure at Randomization (mmHg) [Mean (Standard Deviation); unit: mmHg] | 108 (11) | 107 (9) | 111 (7) | 108 (9) | 103 (8) | 95 (9) | 107 (10)
Diastolic Blood Pressure at Randomization (mmHg) [Mean (Standard Deviation); unit: mmHg] | 62 (7) | 62 (6) | 65 (8) | 65 (8) | 62 (8) | 63 (7) | 63 (7)
DKA at Diagnosis [Count of Participants; unit: Participants]
  Yes | 8 | 7 | 10 | 11 | 11 | 4 | 51
  No | 13 | 13 | 15 | 10 | 7 | 2 | 60
  Missing | 1 | 0 | 0 | 0 | 1 | 0 | 2
Tanner Staging [Count of Participants; unit: Participants] — Tanner stages assess pubertal development in adolescents. Higher stages indicate more advanced pubertal development. Stages are determined by the pubic hair scale for both males and females, the female breast development scale, and the male external genitalia scale.
  Participants
    Group 1 | 6 | 8 | 3 | 4 | 18 | 5 | 44
    Group 2-5 | 16 | 12 | 22 | 17 | 1 | 1 | 69

OUTCOME MEASURES:

1. Primary Outcome: C-peptide Area Under the Curve (AUC)
Description: The primary outcome is the C-peptide in response to a 2-hour MMTT at 52 weeks. C-peptide was measured at 0, 15, 30, 45, 60, 90, and 120 minutes following the start of the mixed meal tolerance test (MMTT). This is summarized as the area under the stimulated C-peptide curve (AUC). AUC is computed using a trapezoidal rule, which is a weighted sum of the C-peptide values over the 120 min.
Time Frame: 52 weeks
Population: 1 participant randomized to Non-HCL and placebo dropped prior to baseline data being collected and was not analyzed. All other participants with at least one available measurement of C-Peptide AUC were included in the analysis model.
Measure: Geometric Mean (Standard Deviation); unit: (pmol/ml)*minutes
Groups:
- HCL and Intensive Management: Participants assigned to HCL group will initially be randomly assigned 1:1 to use either the Tandem t:slim X2 with Control-IQ technology or a Medtronic HCL system (Medtronic 670G 4.0 AHCL (prior to protocol version 5.0) or Medtronic 780G (starting with protocol version 5.0)). This group will receive intensive diabetes management with frequent contacts by study staff with the goal of near-normalization of glucose concentrations.
  [Cohort B participants will not receive study drug. Instead, they will be randomized 2:1 to HCL or non-HCL.] HCL: Hybrid Closed Loop therapy verapamil
- Non-HCL and Standard Care: Participants assigned to non-HCL will receive a Dexcom G6 CGM and diabetes management will follow usual care by their personal diabetes health care provider.
  [Cohort B participants will not receive study drug. Instead, they will be randomized 2:1 to HCL or non-HCL.]
  non-HCL: Usual diabetes care
- Verapamil: Verapamil will be taken orally once per day by participants in Cohort A. A dosing scheme will be followed, using 120mg tablets or 60mg half tablets.
  Whether drug is active or placebo is blinded to both participant and site. [Cohort B participants will not receive study drug. Instead, they will be randomized 2:1 to HCL or non-HCL.]
  verapamil 120mg tablet: verapamil tablet
- Placebo: Placebo will be taken orally once per day by participants in Cohort A. A dosing scheme will be followed, using 120mg tablets or 60mg half tablets.
  Whether drug is active or placebo is blinded to both participant and site.
  [Cohort B participants will not receive study drug. Instead, they will be randomized 2:1 to HCL or non-HCL.]
  placebo: placebo pill manufactured to mimic verapamil 120mg tablet
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
(pmol/ml)*minutes
  Randomization | 0.57 (0.22) | 0.60 (0.18) | 0.66 (0.20) | 0.60 (0.22)
  52 Weeks | 0.45 (0.30) | 0.50 (0.31) | 0.65 (0.31) | 0.44 (0.30)
Statistical Analysis 1: Comparison: HCL and Intensive Management vs Non-HCL and Standard Care; Test type: Superiority; p = 0.89, Mixed Models Analysis; The model included age, days from T1D diagnosis to randomization, and drug group as fixed effects and clinical site as a random effect; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.11 to 0.10] — Mean difference (HCL - Non-HCL) at 52 weeks adjusted for age, days from T1D diagnosis to randomization, RCT drug group, and clinical site
Statistical Analysis 2: Comparison: Verapamil vs Placebo; Test type: Superiority; p = 0.04, Mixed Models Analysis; The model included age, days from T1D diagnosis to randomization, and Intensive group as fixed effects and clinical site as a random effect; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [0.01 to 0.27] — Mean difference (Verapamil - Placebo) at 52 weeks adjusted for age, days from T1D diagnosis to randomization, RCT intensive/standard care group, and clinical site

2. Secondary Outcome: C-peptide AUC
Description: C-peptide AUC between treatment groups. C-peptide was measured at 0, 15, 30, 45, 60, 90, and 120 minutes following the start of the mixed meal tolerance test (MMTT). This is summarized as the area under the stimulated C-peptide curve (AUC). AUC is computed using a trapezoidal rule, which is a weighted sum of the C-peptide values over the 120 min.
Time Frame: 13, 26 and 39 weeks
Population: 1 participant randomized to Non-HCL and placebo dropped prior to baseline data being collected and was not analyzed. All other participants had at least one available measurement of C-peptide AUC and were included in the analysis.
Measure: Geometric Mean (Standard Deviation); unit: (pmol/ml)*minutes
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
(pmol/ml)*minutes
  Randomization | 0.57 (0.22) | 0.60 (0.18) | 0.66 (0.20) | 0.60 (0.22)
  Week 13 | 0.63 (0.23) | 0.69 (0.25) | 0.75 (0.26) | 0.69 (0.23)
  Week 26 | 0.62 (0.28) | 0.63 (0.28) | 0.77 (0.30) | 0.62 (0.25)
  Week 39 | 0.51 (0.30) | 0.57 (0.30) | 0.71 (0.31) | 0.52 (0.28)
Statistical Analysis 1: Comparison: HCL and Intensive Management vs Non-HCL and Standard Care; Test type: Superiority; p = 0.80, Mixed Models Analysis — P-value adjusted for multiplicity using the Benjamini-Hochberg procedure; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.10 to 0.08] — Mean difference (HCL - Non-HCL) at 13 weeks adjusted for age, days from T1D diagnosis to randomization, RCT drug group, and clinical site
Statistical Analysis 2: Comparison: HCL and Intensive Management vs Non-HCL and Standard Care; Test type: Superiority; p = 0.80, Mixed Models Analysis — P-value adjusted for multiplicity using the Benjamini-Hochberg procedure; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.08 to 0.13] — Mean difference (HCL - Non-HCL) at 26 weeks adjusted for age, days from T1D diagnosis to randomization, RCT drug group, and clinical site
Statistical Analysis 3: Comparison: HCL and Intensive Management vs Non-HCL and Standard Care; Test type: Superiority; p = 0.80, Mixed Models Analysis — P-value was adjusted for multiplicity using the Benjamini-Hochberg procedure; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.13 to 0.09] — Mean difference (HCL - Non-HCL) at 39 weeks adjusted for age, days from T1D diagnosis to randomization, RCT drug group, and clinical site
Statistical Analysis 4: Comparison: Verapamil vs Placebo; Test type: Superiority; p = 0.69, Mixed Models Analysis — P-value adjusted for multiplicity using the Benjamini-Hochberg procedure; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.09 to 0.13] — Mean difference (Verapamil - Placebo) at 13 weeks adjusted for age, days from T1D diagnosis to randomization, RCT intensive/standard care group, and clinical site
Statistical Analysis 5: Comparison: Verapamil vs Placebo; Test type: Superiority; p = 0.08, Mixed Models Analysis — P-value was adjusted for multiplicity using the Benjamini-Hochberg procedure; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.02 to 0.25] — Mean difference (Verapamil - Placebo) at 26 weeks adjusted for age, days from T1D diagnosis to randomization, RCT intensive/standard care group, and clinical site
Statistical Analysis 6: Comparison: Verapamil vs Placebo; Test type: Superiority; p = 0.08, Mixed Models Analysis — P-value adjusted for multiplicity using the Benjamini-Hochberg procedure; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.01 to 0.28] — Mean difference (Verapamil - Placebo) at 39 weeks adjusted for age, days from T1D diagnosis to randomization, RCT intensive/standard care group, and clinical site

3. Secondary Outcome: Peak C-peptide
Description: Maximum of all C-peptide values during the MMTT
Time Frame: 13, 26, 39 weeks and 52 weeks
Population: 1 participant randomized to Non-HCL and placebo dropped prior to baseline data being collected and was excluded from the analyses.
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
pmol/mL
  Randomization | 0.72 (0.25) | 0.78 (0.23) | 0.96 (0.30) | 0.89 (0.27)
  13 Weeks | 0.81 (0.27) | 0.87 (0.29) | 0.84 (0.24) | 0.78 (0.27)
  26 Weeks | 0.78 (0.34) | 0.76 (0.33) | 0.97 (0.35) | 0.76 (0.30)
  39 Weeks | 0.65 (0.35) | 0.69 (0.35) | 0.89 (0.36) | 0.63 (0.32)
  52 Weeks | 0.56 (0.36) | 0.62 (0.37) | 0.83 (0.37) | 0.55 (0.34)

4. Secondary Outcome: Number of Participants With a Peak C-peptide >= 0.2 Pmol/ml
Description: Percentage where maximum of all C-peptide values during the MMTT >= 0.2 pmol/ml
Time Frame: 13, 26, 39 weeks and 52 weeks
Population: 1 participant in Non-HCL+Placebo group dropped at baseline and was not analyzed. N missing in each group are as follows; HCL (N=1 at baseline, N=3 at 13 weeks, N=4 at 26 weeks, N=4 at 39 weeks, N=2 at 52 weeks); Non-HCL (N=0 at baseline, N=0 at 13 weeks, N=2 at 26 weeks , N=6 at 39 weeks, N=5 at 52 weeks); Verapamil (N=1 at baseline, N=1 at 13 weeks, N=2 at 26 weeks, N=4 at 39 Weeks, N=4 at 52 weeks); Placebo (N=0 at baseline, N=1 at 13 weeks, N=3 at 26 weeks, N=3 at 39 weeks, N=2 at 52 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
Participants
  Randomization: number analyzed (Participants) | 60 | 51 | 46 | 40
  Randomization | 60 | 51 | 46 | 40
  13 Weeks: number analyzed (Participants) | 58 | 51 | 46 | 39
  13 Weeks | 58 | 50 | 45 | 39
  26 Weeks: number analyzed (Participants) | 57 | 49 | 45 | 37
  26 Weeks | 56 | 47 | 44 | 37
  39 Weeks: number analyzed (Participants) | 57 | 45 | 43 | 37
  39 Weeks | 49 | 38 | 41 | 31
  52 Weeks: number analyzed (Participants) | 59 | 46 | 43 | 38
  52 Weeks | 45 | 36 | 41 | 27

5. Secondary Outcome: CGM Mean Glucose
Description: Mean glucose between treatment groups
Time Frame: 6, 13, 26, 39 weeks and 52 weeks
Population: 1 participant in the Non-HCL+Placebo group dropped at the randomization visit and was not analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
mg/dL
  6 Weeks | 129 (12) | 139 (29) | 131 (23) | 132 (22)
  13 Weeks | 132 (15) | 140 (26) | 134 (22) | 134 (22)
  26 Weeks | 135 (17) | 152 (35) | 138 (32) | 144 (27)
  39 Weeks | 140 (19) | 161 (36) | 141 (23) | 155 (38)
  52 Weeks | 145 (19) | 167 (42) | 151 (27) | 159 (41)
Statistical Analysis 1: Comparison: HCL and Intensive Management vs Non-HCL and Standard Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -25, 95% CI 2-sided [-37 to -14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Verapamil vs Placebo; Test type: Superiority; p = 0.74, Mixed Models Analysis; Mean Difference (Final Values) = -4, 95% CI 2-sided [-25 to 16] — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Percentage of CGM Time in Range (70-180 mg/dL)
Description: CGM sensor glucose values from 70 to 180 mg/dL between treatment groups
Time Frame: 6, 13, 26, 39 weeks and 52 weeks
Population: 1 participant in the Non-HCL+Placebo group dropped at the randomization visit and was not analyzed.
Measure: Mean (Standard Deviation); unit: Percent of Time
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
Percent of Time
  6 Weeks | 86 (8) | 84 (9) | 85 (15) | 84 (13)
  13 Weeks | 84 (9) | 79 (16) | 83 (15) | 84 (13)
  26 Weeks | 83 (10) | 73 (20) | 81 (17) | 78 (17)
  39 Weeks | 80 (11) | 68 (21) | 80 (15) | 72 (20)
  52 Weeks | 78 (11) | 64 (22) | 74 (18) | 70 (21)
Statistical Analysis 1: Comparison: HCL and Intensive Management vs Non-HCL and Standard Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 16, 95% CI 2-sided [10 to 22] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Verapamil vs Placebo; Test type: Superiority; p = 0.74, Mixed Models Analysis; Mean Difference (Final Values) = 2, 95% CI 2-sided [-9 to 13] — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: Percentage of CGM Time in Range 70-140 mg/dL
Description: Percentage of CGM sensor glucose values from 70 to 140 mg/dL between treatment groups
Time Frame: 6, 13, 26, 39 weeks and 52 weeks
Population: 1 participant in the Non-HCL+Placebo group dropped at the randomization visit and was not analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
Percentage of Time
  6 Weeks | 69 (11) | 60 (22) | 67 (19) | 66 (18)
  13 Weeks | 67 (13) | 59 (22) | 65 (19) | 65 (19)
  26 Weeks | 64 (13) | 51 (21) | 61 (20) | 57 (19)
  39 Weeks | 60 (14) | 46 (21) | 58 (19) | 51 (20)
  52 Weeks | 56 (13) | 43 (21) | 51 (19) | 49 (21)
Statistical Analysis 1: Comparison: HCL and Intensive Management vs Non-HCL and Standard Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 16, 95% CI 2-sided [10 to 22] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Verapamil vs Placebo; Test type: Superiority; p = 0.95, Mixed Models Analysis; Mean Difference (Final Values) = 0, 95% CI 2-sided [-8 to 14] — [estimate comment as in outcome 1, analysis 2]

8. Secondary Outcome: Number of Participants With CGM Time in Range 70-180 mg/dL >=70% at 52 Weeks
Description: Percentage of patients with >=70% sensor glucose values from 70 to 180 mg/dL between treatment groups
Time Frame: 52 Weeks
Population: N missing in each group are as follows; HCL (N=2 at 52 weeks); Non-HCL (N=4 at 52 weeks); Verapamil (N=3 at 52 weeks); Placebo (N=3 at 52 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 59 | 47 | 44 | 37
Participants | 46 | 22 | 30 | 23
Statistical Analysis 1: Comparison: HCL and Intensive Management vs Non-HCL and Standard Care; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 0.38, 95% CI 2-sided [0.21 to 0.53]
Statistical Analysis 2: Comparison: Verapamil vs Placebo; Test type: Superiority; p = 0.79, Regression, Logistic; Risk Difference (RD) = 0.03, 95% CI 2-sided [-0.26 to 0.32]

9. Secondary Outcome: Percentage of CGM Time >140 mg/dL
Description: CGM sensor glucose values >140 mg/dL between treatment groups
Time Frame: 6, 13, 26, 39 weeks and 52 weeks
Population: 1 participant in Non-HCL+Placebo group dropped at baseline and was not analyzed.
Measure: Mean (Standard Deviation); unit: Percent of Time
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
Percent of Time
  6 Weeks | 29 (11) | 38 (23) | 32 (19) | 32 (18)
  13 Weeks | 32 (13) | 40 (22) | 34 (19) | 33 (20)
  26 Weeks | 34 (13) | 47 (22) | 36 (20) | 41 (20)
  39 Weeks | 38 (14) | 53 (21) | 40 (19) | 47 (21)
  52 Weeks | 42 (14) | 56 (22) | 47 (19) | 49 (22)

10. Secondary Outcome: Percentage of CGM Time >180 mg/dL
Description: CGM sensor glucose values >180 mg/dL between treatment groups
Time Frame: 6, 13, 26, 39 weeks and 52 weeks
Population: 1 participant in Non-HCL+Placebo group dropped at baseline and was not analyzed.
Measure: Mean (Standard Deviation); unit: Percent of Time
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
Percent of Time
  6 Weeks | 12 (8) | 19 (19) | 13 (15) | 14 (14)
  13 Weeks | 14 (9) | 19 (17) | 15 (15) | 15 (14)
  26 Weeks | 15 (10) | 25 (20) | 17 (17) | 21 (18)
  39 Weeks | 18 (11) | 30 (21) | 19 (15) | 26 (21)
  52 Weeks | 20 (11) | 34 (22) | 25 (18) | 28 (21)
Statistical Analysis 1: Comparison: HCL and Intensive Management vs Non-HCL and Standard Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -16, 95% CI 2-sided [-22 to -9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Verapamil vs Placebo; Test type: Superiority; p = 0.74, Mixed Models Analysis; Mean Difference (Final Values) = -2, 95% CI 2-sided [-13 to 9] — Mean difference at 52 weeks (verapamil - placebo) adjusted for age, days from T1D diagnosis to randomization, RCT intensive/standard care group, and clinical site

11. Secondary Outcome: Percentage of CGM Time >250 mg/dL
Description: Percentage of CGM sensor glucose values >250 mg/dL between treatment groups
Time Frame: 6, 13, 26, 39 weeks and 52 weeks
Population: 1 participant in Non-HCL+Placebo group dropped at baseline and was not analyzed.
Measure: Mean (Standard Deviation); unit: Percent of Time
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
Percent of Time
  6 Weeks | 1 (2) | 3 (4) | 1 (1) | 2 (3)
  13 Weeks | 2 (3) | 3 (4) | 2 (2) | 2 (3)
  26 Weeks | 2 (3) | 6 (8) | 2 (3) | 4 (6)
  39 Weeks | 3 (3) | 9 (12) | 3 (4) | 7 (9)
  52 Weeks | 4 (4) | 10 (13) | 5 (6) | 8 (10)
Statistical Analysis 1: Comparison: HCL and Intensive Management vs Non-HCL and Standard Care; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -4, 95% CI 2-sided [-7 to -1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Verapamil vs Placebo; Test type: Superiority; p = 0.74, Mixed Models Analysis; Mean Difference (Final Values) = -1, 95% CI 2-sided [-6 to 4] — [estimate comment as in outcome 1, analysis 2]

12. Secondary Outcome: Percentage of CGM Time <54 mg/dL
Description: Percentage of CGM sensor glucose values <54 mg/dL between treatment groups
Time Frame: 6, 13, 26, 39 weeks and 52 weeks
Population: 1 participant in Non-HCL+Placebo group dropped at baseline and was not analyzed.
Measure: Mean (Standard Error); unit: Percent of Time
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
Percent of Time
  6 Weeks | 0.22 (0.22) | 0.11 (0.13) | 0.14 (0.16) | 0.16 (0.16)
  13 Weeks | 0.23 (0.21) | 0.12 (0.16) | 0.19 (0.20) | 0.16 (0.19)
  26 Weeks | 0.25 (0.25) | 0.10 (0.11) | 0.22 (0.25) | 0.14 (0.18)
  39 Weeks | 0.32 (0.34) | 0.16 (0.20) | 0.21 (0.27) | 0.26 (0.27)
  52 Weeks | 0.29 (0.34) | 0.18 (0.21) | 0.20 (0.24) | 0.24 (0.26)
Statistical Analysis 1: Comparison: HCL and Intensive Management vs Non-HCL and Standard Care; Test type: Superiority; p = 0.23, Regression, Linear; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.04 to 0.17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Verapamil vs Placebo; Test type: Superiority; p = 0.79, Regression, Linear; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.0 to 0.6] — [estimate comment as in outcome 1, analysis 2]

13. Secondary Outcome: Percentage of CGM Time <70 mg/dL
Description: Percentage of CGM sensor glucose values <70 mg/dL between treatment groups
Time Frame: 6, 13, 26, 39 weeks and 52 weeks
Population: 1 participant in Non-HCL+Placebo group dropped at baseline and was not analyzed.
Measure: Mean (Standard Deviation); unit: Percent of Time
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
Percent of Time
  6 Weeks | 1.7 (1.0) | 1.5 (1.6) | 1.5 (1.5) | 1.7 (1.6)
  13 Weeks | 1.6 (1.2) | 1.2 (1.1) | 1.4 (0.9) | 1.4 (1.5)
  26 Weeks | 1.9 (1.1) | 1.2 (1.0) | 1.6 (1.4) | 1.4 (1.2)
  39 Weeks | 2.0 (1.3) | 1.2 (1.3) | 1.5 (1.4) | 1.7 (1.6)
  52 Weeks | 1.8 (1.2) | 1.4 (1.4) | 1.3 (1.2) | 1.6 (1.3)
Statistical Analysis 1: Comparison: HCL and Intensive Management vs Non-HCL and Standard Care; Test type: Superiority; p = 0.39, Regression, Linear; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.3 to 0.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Verapamil vs Placebo; Test type: Superiority; p = 0.74, Regression, Linear; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.0 to 0.6] — [estimate comment as in outcome 1, analysis 2]

14. Secondary Outcome: CGM Coefficient of Variation
Description: Coefficient of variation between treatment groups. Calculated as the standard deviation of CGM glucose values divided by the mean of CGM glucose values.
Time Frame: 6, 13, 26, 39 weeks and 52 weeks
Population: 1 participant in Non-HCL+Placebo group dropped at baseline and was not analyzed.
Measure: Mean (Standard Deviation); unit: Coefficient of Variation Percentage
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
Coefficient of Variation Percentage
  6 Weeks | 31 (5) | 30 (6) | 28 (5) | 30 (6)
  13 Weeks | 31 (6) | 30 (7) | 29 (6) | 29 (6)
  26 Weeks | 32 (5) | 32 (6) | 30 (6) | 31 (5)
  39 Weeks | 34 (6) | 33 (6) | 31 (6) | 33 (5)
  52 Weeks | 34 (6) | 33 (5) | 32 (6) | 33 (5)

15. Secondary Outcome: HbA1c
Description: HbA1c between treatment groups
Time Frame: 13, 26, 39 weeks and 52 weeks
Population: 1 participant in Non-HCL+Placebo group dropped at baseline and was not analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of Glycosylated Hemoglobin
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
Percentage of Glycosylated Hemoglobin
  Randomization | 10.3 (1.3) | 10.2 (1.6) | 10.3 (1.7) | 10.2 (1.2)
  13 Weeks | 6.4 (0.5) | 6.5 (0.9) | 6.3 (0.8) | 6.4 (0.6)
  26 Weeks | 6.4 (0.6) | 6.6 (1.0) | 6.3 (0.9) | 6.5 (0.8)
  39 Weeks | 6.6 (0.7) | 7.0 (1.2) | 6.4 (0.9) | 7.0 (1.1)
  52 Weeks | 6.5 (0.7) | 7.1 (1.3) | 6.6 (1.0) | 6.9 (1.2)
Statistical Analysis 1: Comparison: HCL and Intensive Management vs Non-HCL and Standard Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.1 to -0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Verapamil vs Placebo; Test type: Superiority; p = 0.65, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.0 to 0.4] — [estimate comment as in outcome 1, analysis 2]

16. Secondary Outcome: Number of Participants With HbA1c <7.0%
Description: Percentage of participants with HbA1c < 7.0% between treatment groups
Time Frame: 13, 26, 39 weeks and 52 weeks
Population: 1 participant in Non-HCL+Placebo group dropped at baseline and was not analyzed. N missing in each group are as follows; HCL (N=1 at baseline, N=3 at 13 weeks, N=4 at 26 weeks, N=2 at 39 weeks, N=2 at 52 weeks); Non-HCL (N=0 at baseline, N=0 at 13 weeks, N=2 at 26 weeks , N=5 at 39 weeks, N=3 at 52 weeks); Verapamil (N=0 at baseline, N=0 at 13 weeks, N=2 at 26 weeks, N=4 at 39 Weeks, N=4 at 52 weeks); Placebo (N=1 at baseline, N=1 at 13 weeks, N=3 at 26 weeks, N=1 at 39 weeks, N=1 at 52 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
Participants
  Randomization: number analyzed (Participants) | 60 | 51 | 47 | 39
  Randomization | 2 | 1 | 3 | 0
  13 Weeks: number analyzed (Participants) | 58 | 51 | 47 | 39
  13 Weeks | 48 | 36 | 38 | 32
  26 Weeks: number analyzed (Participants) | 57 | 49 | 45 | 37
  26 Weeks | 45 | 31 | 37 | 25
  39 Weeks: number analyzed (Participants) | 59 | 46 | 43 | 39
  39 Weeks | 44 | 23 | 33 | 22
  52 Weeks: number analyzed (Participants) | 59 | 48 | 43 | 39
  52 Weeks | 42 | 26 | 32 | 23

17. Secondary Outcome: Number of Participants With HbA1c <6.5%
Description: Percentage of participants with HbA1c < 6.5% between treatment groups
Time Frame: 13, 26, 39 weeks and 52 weeks
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
Participants
  Randomization: number analyzed (Participants) | 60 | 51 | 47 | 39
  Randomization | 0 | 0 | 0 | 0
  13 Weeks: number analyzed (Participants) | 58 | 51 | 47 | 39
  13 Weeks | 27 | 24 | 27 | 20
  26 Weeks: number analyzed (Participants) | 57 | 49 | 45 | 37
  26 Weeks | 37 | 23 | 31 | 22
  39 Weeks: number analyzed (Participants) | 59 | 46 | 43 | 39
  39 Weeks | 33 | 20 | 30 | 18
  52 Weeks: number analyzed (Participants) | 59 | 48 | 43 | 39
  52 Weeks | 28 | 19 | 25 | 18

18. Secondary Outcome: Total Daily Insulin Per kg
Description: Total daily insulin per kg between treatment groups
Time Frame: 6, 13, 26, 39 weeks and 52 weeks
Population: 1 participant in Non-HCL+Placebo group dropped at baseline and was not analyzed.
Measure: Mean (Standard Deviation); unit: U/kg/day
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
U/kg/day
  Randomization | 0.68 (0.28) | 0.66 (0.30) | 0.74 (0.29) | 0.64 (0.27)
  6 Weeks | 0.54 (0.26) | 0.55 (0.33) | 0.55 (0.33) | 0.54 (0.28)
  13 Weeks | 0.51 (0.23) | 0.53 (0.25) | 0.54 (0.25) | 0.54 (0.26)
  26 Weeks | 0.61 (0.28) | 0.53 (0.23) | 0.57 (0.28) | 0.58 (0.29)
  39 Weeks | 0.68 (0.32) | 0.58 (0.27) | 0.59 (0.29) | 0.66 (0.32)
  52 Weeks | 0.74 (0.32) | 0.64 (0.25) | 0.65 (0.26) | 0.74 (0.34)
Statistical Analysis 1: Comparison: HCL and Intensive Management vs Non-HCL and Standard Care; Test type: Superiority; p = 0.07, Mixed Models Analysis; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.01 to 0.20] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Verapamil vs Placebo; Test type: Superiority; p = 0.52, Mixed Models Analysis; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.30 to 0.05] — [estimate comment as in outcome 1, analysis 2]

19. Secondary Outcome: Basal:Bolus Ratio
Description: Ratio of basal:bolus insulin between treatment groups
Time Frame: 6, 13, 26, 39 weeks and 52 weeks
Population: 1 participant in Non-HCL+Placebo group dropped at baseline and was not analyzed.
Measure: Number; unit: Daily Basal/Bolus Ratio
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 40
Daily Basal/Bolus Ratio
  Randomization | 0.96 | 1.0 | 1.1 | 1.1
  6 Weeks | 0.61 | 1.1 | 0.89 | 0.85
  13 Weeks | 0.61 | 1 | 0.89 | 0.82
  26 Weeks | 0.59 | 0.85 | 0.72 | 0.75
  39 Weeks | 0.67 | 0.72 | 0.75 | 0.72
  52 Weeks | 0.69 | 0.75 | 0.82 | 0.72

20. Secondary Outcome: Severe Hypoglycemia
Description: Frequency of episodes of severe hypoglycemia between treatment groups
Time Frame: 52 weeks
Measure: Number; unit: Number of Severe Hypoglycemic Events
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 41
Number of Severe Hypoglycemic Events | 1 | 1 | 1 | 1

21. Secondary Outcome: DKA
Description: Frequency of episodes of DKA between treatment groups
Time Frame: 52 weeks
Measure: Number; unit: Number of DKA Events
Arm/Group | HCL and Intensive Management | Non-HCL and Standard Care | Verapamil | Placebo
Number analyzed (Participants) | 61 | 51 | 47 | 41
Number of DKA Events | 1 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data where collected during the 52 week RCT phase.
Arm/Group | HCL and Verapamil | HCL and Placebo | Non-HCL and Verapamil | Non-HCL and Placebo | HCL Only | Non-HCL Only
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20 | 0/25 | 0/21 | 0/19 | 0/6
Serious Adverse Events (participants affected / at risk) | 3/22 | 1/20 | 1/25 | 3/21 | 1/19 | 0/6
Other Adverse Events (participants affected / at risk) | 20/22 | 16/20 | 19/25 | 14/21 | 18/19 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCL and Verapamil (N=22) | HCL and Placebo (N=20) | Non-HCL and Verapamil (N=25) | Non-HCL and Placebo (N=21) | HCL Only (N=19) | Non-HCL Only (N=6)
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic Ketoacidosis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCL and Verapamil (N=22) | HCL and Placebo (N=20) | Non-HCL and Verapamil (N=25) | Non-HCL and Placebo (N=21) | HCL Only (N=19) | Non-HCL Only (N=6)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swollen Glands (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
2nd Degree Heart Block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
1st Degree Heart Block (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Premature Ventricular Contractions (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Infection (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis Externa (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis Media Acute (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain in Ear (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Endocrine disorders) | 3 (6) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acid Indegestion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bloody Stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Celiac Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach Virus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth Infection (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upset Stomach (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Catheter Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 5 (6) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Swelling of Feet (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy NOS (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hives (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vitiligo (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 3 (3) | 4 (4) | 6 (7) | 3 (3) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tinea Pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Syndrome (Infections and infestations) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Animal Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated Liver Enzymes (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Heart Murmur (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal Weight Gain (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 1 (2) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arm Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leg Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leg Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in Elbow (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sprained Ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temporomandibular Joint Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 3 (4) | 1 (1) | 4 (4) | 3 (7) | 0 (0)
Numbness in Feet (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pre-syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tingling Sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasovagal Attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adjustment Disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Panic Attack (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Streptococcal Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bruise (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ingrown toe nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin Abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Bacterial Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Disorder NOS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Tinea Corporis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Benign Essential Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT04233034/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT04233034/SAP_001.pdf